CLINICAL TRIAL: NCT01843595
Title: Efficacy Trial of the REFIT (Rethinking Eating and FITness) Weight Loss Intervention for Men
Brief Title: Rethinking Eating and FITness for Men
Acronym: REFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-1548
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-09

CONDITIONS: Weight Loss; Overweight
MeSH Terms: conditions — Weight Loss; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- REFIT Intervention (Experimental): This arm will receive the REFIT intervention immediately after randomization.
  Interventions: Behavioral: REFIT Intervention
- Wait-list control (No Intervention): This arm will receive a modified version of the REFIT program after the 6-month assessment.

INTERVENTIONS:
Behavioral: REFIT Intervention — The intervention will include 2 face-to-face group meetings, weekly check-in sessions, weekly tailored feedback, and weekly lessons focused on specific weight loss behaviors. All participants will be encouraged increase their physical activity to approximately 250 minutes of moderate to vigorous physical activity per week.
  Arms: REFIT Intervention

SUMMARY:
The purpose of this study is to test the effect of a new three-month behavioral weight loss program among adult men. Weight will be measured at three and six months post randomization. The intervention will be compared to a wait-list control group. Participants will be 112 overweight and obese men (18-65) living in the Chapel Hill/Raleigh/Durham area. The behavioral intervention tested will be delivered online with two face-to-face group meetings. Intervention content will be delivered via email and online. It is hypothesized that men randomized to the REFIT intervention will lose more weight at 3 months than men randomized to the wait-list group.

DETAILED DESCRIPTION:
Obesity is one of the greatest threats to modern public health. It is associated with negative physical and mental health outcomes as well as increased healthcare expenditures. Throughout the time period that the prevalence of overweight and obesity have been monitored in the United States, men have consistently been more likely than women to be overweight and; conversely, women have been more likely to be obese. Recent trends suggest that this situation may be changing. Over the past decade, the prevalence of obesity has increased among men while it has stabilized among women. For the first time, men and women have near equal rates of obesity where approximately 35.7% of American adults are classified as obese; meanwhile, men continue to be more overweight than women.

The epidemiological trends have lead to a focus on creating weight loss programs that can aid overweight and obese adults in losing excess weight. Behavioral interventions for obesity have demonstrated the ability to produce weight losses of approximately 5-10% of initial body weight. These weight losses have been associated with decreased risk for type II diabetes, reduced blood pressure, and improvement in mental health outcomes. Unfortunately, men typically do not take advantage of such programs. Across multiple literature reviews, men consistently make up approximately 27% of study samples. This has lead to a situation where researchers have little information about how to enroll men in weight loss programs and what kind of programs are of interest to men. In order to combat the increased obesity in men and help them to avoid the negative consequences of obesity, it is important to help overweight and obese men change their eating and physical activity habits within the context of organized weight loss programs.

The REFIT (Rethinking Eating and FITness) intervention is an intervention developed to address men's needs for weight loss while balancing their need to perform behaviors which are seen as masculine. Men typically eat a diet that is associated with weight gain rather than weight loss. The REFIT intervention will focus on changing eating and exercise behaviors within a structured weight loss program that will allow men to maintain their autonomy. Autonomy is a central characteristic of enacted masculinity and has been described in qualitative research as a necessary aspect of a weight loss program for men. The intervention will focus on encouraging changes in eating and activity through increasing self-efficacy, autonomous motivation, outcome expectancies, and self-regulation for weight loss behaviors. The development of this intervention has been guided by qualitative research focused on what men want and need from weight loss programs as well as previous research focused on weight loss among both men and women. The approach to be used in the REFIT intervention is innovative as a combination of the "small changes" approach that has been used in weight gain prevention as well as the client centered deficit approaches used by Lutes and colleagues and Sbrocco and colleagues in weight loss programs.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-65 years of age
* Body mass index between 25-40 kg/m²
* Able to access the Internet at least twice weekly
* Able to read and write in English
* Able to attend two group sessions at the UNC Weight Research Program clinic site

Exclusion Criteria:

* Lost more than 10 pounds over the last 6 months
* Currently participating in another weight loss program
* Report a diagnosis of schizophrenia, bipolar disorder, or substance abuse, or depression leading to hospitalization during the previous year
* Currently being treated for cancer
* Unable to exercise safely (as defined as endorsement of items 1-4 of the Physical Activity Readiness Questionnaire)
* Heavy use or abuse of alcohol (as defined as a score of 8 or higher on the Alcohol Disorders Identification Test)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in weight from baseline to 3 months | Baseline, 3 months
  Weight will be collected at baseline and 3 months at the UNC Weight Research Program Center and measured to the nearest 0.1 kg using a digital Tanita scale that will be calibrated routinely. Participants will weigh-in wearing shorts and no shoes.

SECONDARY OUTCOMES:
Change in weight from baseline to 6 months | Baseline, 6 months
  Weight will be collected at baseline and 6 months at the UNC Weight Research Program Center and measured to the nearest 0.1 kg using a digital Tanita scale that will be calibrated routinely. Participants will weigh-in wearing shorts and no shoes.
Change in caloric intake between baseline and 3 months | Baseline, 3 months
  Caloric intake will be assessed at baseline and 3 months using the online Automated Self-Administered 24-hour recall tool created by the National Cancer Institute.
Change in physical activity between baseline and 3 months | Baseline, 3 months
  Energy expenditure from exercise will be assessed at baseline and 3 months via the Paffenbarger Exercise Habits Questionnaire.
Self-efficacy for weight loss behaviors at 3 months | 3 months
  Self-efficacy for eating behaviors related to weight control will be measured at 3 months using the Weight Efficacy Lifestyle Questionnaire.
Motivation for healthy eating at 3 months | 3 months
  Motivation for healthy eating will be measured at 3 months using the Treatment Self-Regulation Questionnaire for Healthy Eating.
Motivation for Physical Activity at 3 months | 3 months
  Motivation for physical activity will be measured at 3 months using the Treatment Self-Regulation Questionnaire for Physical Activity.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Crane, MA, Principal Investigator — University of North Carolina, Chapel Hill; Deborah F. Tate, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Crane MM, Ward DS, Lutes LD, Bowling JM, Tate DF. Theoretical and Behavioral Mediators of a Weight Loss Intervention for Men. Ann Behav Med. 2016 Jun;50(3):460-70. doi: 10.1007/s12160-016-9774-z. PMID 26842133